CLINICAL TRIAL: NCT06865521
Title: Safety and Feasibility of Akkermansia Probiotics Combined With Anti-PD-1 Monoclonal Antibody in MSS/pMMR Advanced Colorectal Cancer
Brief Title: Akkermansia Probiotics Plus Anti-PD-1 Monoclonal Antibody in MSS/pMMR Advanced Colorectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Principal Investigator, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKPP-I 2025-2-21
Record Dates: First submitted 2025-02-21; First posted 2025-03-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Colo-rectal Cancer; PD-1 Inhibitor; Akkermansia Muciniphila
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: anti-PD-1 monoclonal antibody + TKI (TKI, e.g., regorafenib, fruquintinib) treatment / anti-PD-1 monoclonal antibody ± Chemotherapy (etc., CAPEOX, XELIRI) ± Bevacizumab treatment + Akkermansia probiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self control group (Other): According to the inclusion and exclusion criteria, 22 patients will be recruited. After enrollment, patients will receive anti-PD-1 monoclonal antibody + Tyrosine kinase inhibitor (TKI, e.g., regorafenib, fruquintinib) treatment or anti-PD-1 monoclonal antibody ± chemotherapy (etc., CAPEOX [oxaliplatin+capecitabine ], XELIRI [irinotecan+capecitabine ]) ± Bevacizumab treatment (anti-PD-1 monoclonal antibody, chemotherapy, and bevacizumab every 3 weeks, TKI every 4 weeks), along with daily continuous administration of Akkermansia probiotics (Songke, dose: 1 capsule/day, taken with breakfast), until disease progression, intolerable toxicity, or patient withdrawal from the study.
  Interventions: Dietary Supplement: Akkermansia Probiotics

INTERVENTIONS:
Dietary Supplement: Akkermansia Probiotics — After enrollment, patients will receive anti-PD-1 monoclonal antibody + Tyrosine kinase inhibitor (TKI, e.g., regorafenib, fruquintinib) treatment or anti-PD-1 monoclonal antibody ± chemotherapy (etc., CAPEOX [oxaliplatin+capecitabine ], XELIRI [irinotecan+capecitabine ]) ± Bevacizumab treatment (anti-PD-1 monoclonal antibody, chemotherapy, and bevacizumab every 3 weeks, TKI every 4 weeks), along with daily continuous administration of Akkermansia probiotics (Songke, dose: 1 capsule/day, taken with breakfast), until disease progression, intolerable toxicity, or patient withdrawal from the study.

SUMMARY:
The investigators propose to conduct a single-center, single-arm, Phase I clinical study to explore the safety and feasibility of Akkermansia probiotics combined with anti-PD-1 monoclonal antibody in patients with MSS/pMMR advanced colorectal cancer, as well as its impact on gut microbiota and the immune microenvironment.

DETAILED DESCRIPTION:
Safety and Feasibility of Akkermansia Probiotics Combined with Anti-PD-1 Monoclonal Antibody in MSS/pMMR Advanced Colorectal Cancer The investigators propose to conduct a single-center, single-arm, Phase I clinical study to explore the safety and efficacy of Akkermansia probiotics combined with anti-PD-1 monoclonal antibody in patients with MSS/pMMR advanced colorectal cancer, as well as its impact on gut microbiota and the immune microenvironment.

Inclusion Criteria:

* Age 18-75 years
* ECOG performance status score of 0-2
* Histopathologically confirmed colorectal cancer; tumor tissue immunohistochemistry or genetic testing showing pMMR or MSS/MSI-L type
* Metastatic colorectal adenocarcinoma that has failed standard treatments (including irinotecan, oxaliplatin, fluorouracil, bevacizumab, cetuximab, etc.)
* No prior use of immunotherapy (such as immune checkpoint inhibitors, adoptive cell immunotherapy, etc.)
* At least one evaluable lesion according to RECIST version 1.1 criteria
* No intestinal obstruction and good oral compliance
* Adequate bone marrow, liver, and kidney function to receive treatment
* Signed informed consent

Exclusion Criteria:

* History of allergic diseases, severe drug allergies, or known allergies to probiotic drugs
* Use of antibiotics or probiotic drugs/health products within the last 3 months
* History of other malignancies with a disease-free interval of less than 5 years (except for cured basal cell carcinoma of the skin, cured cervical carcinoma in situ, and gastrointestinal tumors cured by endoscopic mucosal resection)
* Presence of any active autoimmune disease or history of autoimmune disease
* Current use of immunosuppressants or hormone therapy, continued within 2 weeks prior to enrollment
* Concurrent severe infections
* Congenital or acquired immune deficiency, or active hepatitis
* Concurrent severe complications

Intervention Strategy:

According to the inclusion and exclusion criteria, 22 patients will be recruited. After enrollment, patients will receive anti-PD-1 monoclonal antibody + Tyrosine kinase inhibitor (TKI, e.g., regorafenib, fruquintinib) treatment or anti-PD-1 monoclonal antibody ± chemotherapy (etc., CAPEOX [oxaliplatin+capecitabine ], XELIRI [irinotecan+capecitabine ]) ± Bevacizumab treatment (anti-PD-1 monoclonal antibody, chemotherapy, and bevacizumab every 3 weeks, TKI every 4 weeks), along with daily continuous administration of Akkermansia probiotics (Songke, dose: 1 capsule/day, taken with breakfast), until disease progression, intolerable toxicity, or patient withdrawal from the study.

Primary Observation Indicators:

Gastrointestinal adverse reactions, including nausea, vomiting, diarrhea, abdominal pain, etc., and quality of life assessment.

Secondary Indicators:

* Objective Response Rate (ORR): The proportion of patients with a measurable reduction in tumor burden (defined by standardized criteria such as RECIST 1.1) who achieve either a complete response (CR) or a partial response (PR) during the course of treatment.
* Progression-Free Survival (PFS) ：The length of time during and after treatment that a patient lives with the disease without it getting worse. It is typically measured from the start of treatment (or randomization in a clinical trial) until the date of disease progression or death from any cause, whichever occurs first.
* Overall Survival (OS): The duration from the start of treatment (or randomization in a clinical trial) until death from any cause.

Exploratory Indicators:

Changes in the immune microenvironment such as proportions of common immune cells in peripheral blood (CD3+, CD4+, CD8+ T cells, macrophages, dendritic cells, MDSC, etc.), fetal Akkermansia abundance, gut microbiota, and metabolomics.

1. Evaluation of the Safety and Efficacy of Combined Treatment (Incomplete) Quality of life of enrolled patients will be assessed using the EORTC QLQ-C30 scale. Baseline and every 3 weeks, hematological tests (blood routine, liver and kidney function, electrolytes, myocardial markers, thyroid function, etc.) will be conducted to assess bone marrow, liver, and kidney function for adverse reactions. Baseline and every 2 months, imaging (chest and abdominal enhanced CT) will be performed to evaluate tumor efficacy. Patients will be followed up every 2 weeks after enrollment, with follow-up content including treatment tolerance, adverse reactions, survival status, etc.
2. Exploration of the Impact of Akkermansia on Gut Microbiota and the Immune Microenvironment in Colorectal Cancer Patients Treated with Anti-PD-1 Monoclonal Antibody (Incomplete) Baseline and every 3 weeks after enrollment, stool and peripheral blood samples will be collected to detect changes in fecal Akkermansia abundance and gut microbiota, as well as changes in the immune microenvironment such as proportions of common immune cells in peripheral blood (CD3+, CD4+, CD8+ T cells, macrophages, dendritic cells, MDSC, etc.).

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-75 years

  * ECOG performance status score of 0-2
  * Histopathologically confirmed colorectal cancer; tumor tissue immunohistochemistry or genetic testing showing pMMR or MSS/MSI-L type
  * Metastatic colorectal adenocarcinoma that has failed standard treatments (including irinotecan, oxaliplatin, fluorouracil, bevacizumab, cetuximab, etc.)
  * No prior use of immunotherapy (such as immune checkpoint inhibitors, adoptive cell immunotherapy, etc.)
  * At least one evaluable lesion according to RECIST version 1.1 criteria
  * No intestinal obstruction and good oral compliance
  * Adequate bone marrow, liver, and kidney function to receive treatment
  * Signed informed consent

Exclusion Criteria:

* • History of allergic diseases, severe drug allergies, or known allergies to probiotic drugs

  * Use of antibiotics or probiotic drugs/health products within the last 3 months
  * History of other malignancies with a disease-free interval of less than 5 years (except for cured basal cell carcinoma of the skin, cured cervical carcinoma in situ, and gastrointestinal tumors cured by endoscopic mucosal resection)
  * Presence of any active autoimmune disease or history of autoimmune disease
  * Current use of immunosuppressants or hormone therapy, continued within 2 weeks prior to enrollment
  * Concurrent severe infections
  * Congenital or acquired immune deficiency, or active hepatitis
  * Concurrent severe complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2027-03-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From enrollment to one months after study exit
  Physical Symptoms (Nausea, vomiting, headache, dizziness, fatigue, rash, itching, pain, etc); Laboratory Abnormalities: (Abnormal blood test results); Clinical Signs (ever, swelling, high blood pressure, low blood pressure, rapid heart rate, etc); Worsening of Pre-existing Conditions (xacerbation of a pre-existing disease or medical condition); New Medical Conditions (Development of new diseases or disorders that were not present before treatment); Psychological Effects (Anxiety, depression, insomnia, confusion, etc).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 months
  The proportion of patients with a measurable reduction in tumor burden (defined by standardized criteria such as RECIST 1.1) who achieve either a complete response (CR) or a partial response (PR) during the course of treatment.
Relative abundance of Akkermansia muciniphila (AKK) in fecal samples measured by qPCR | Through study completion, an average of 2 months
Quantitative analysis of peripheral blood immune cell subsets (CD8+ T cells, DC subtypes, MDSCs,, etc.) by flow cytometr | Through study completion, an average of 2 months
Serum cytokine profiling (IFN-γ, TNF-α, etc.) by ELISA | Through study completion, an average of 2 months
Changes in gut microbiome composition measured by 16S rRNA gene sequencing analysis | Through study completion, an average of 2 months
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The length of time during and after treatment that a patient lives with the disease without it getting worse.
Overall Survival (OS) | Up to 36 months
  The duration from the start of treatment (or randomization in a clinical trial) until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Cancer, West China Hospital, Chengdu, Sichuan, China